CLINICAL TRIAL: NCT03022955
Title: Effects of Cocoa Solids on Gastrointestinal Transit, Postprandial Sensation and Gastrointestinal Well-being: a Randomized, Controlled Trial in Healthy Volunteers
Brief Title: Effects of Cocoa on Gastrointestinal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Chocolate Study
Record Dates: First submitted 2017-01-10; First posted 2017-01-18 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Gastrointestinal and Digestive Disorder
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dark chocolate: FDG-PET (Active Comparator): 100 g dark chocolate bar (70% cocoa solids (~500kcal, ~50% fat)) will be consumed with radio-opaque markers on three consecutive days. On the third day chocolate ingestion will be followed by measurements of postprandial brain activity and colonic transit using chocolate: fluorodeoxyglucose Positron Emission Tomography (FDG-PET)
  Interventions: Dietary Supplement: Dark chocolate bar
- Dark chocolate: Physiological Measurement (Active Comparator): 150 g dark chocolate mousse (~500kcal, ~50% fat) labelled with 13C-lactose-ureide and technetium (99Tc) will be consumed to assess gastric emptying and oro-caecal transit time by scintigraphy.
  Interventions: Dietary Supplement: Dark chocolate mousse
- White chocolate: FDG-PET (Placebo Comparator): 100 g white chocolate bar (0% cocoa solids (~500kcal, 50% fat) will be consumed with radio-opaque markers on three consecutive days. On the third day chocolate ingestion will be followed by measurements of postprandial brain activity and colonic transit using FDG-Positron Emission Tomography.
  Interventions: Dietary Supplement: White chocolate bar
- White chocolate: Physiological Measurement (Placebo Comparator): 150 g white chocolate mousse (~500kcal, ~50% fat) labelled with 13C-lactose-ureide and technetium (99Tc) will be consumed to assess gastric emptying and oro-caecal transit time by scintigraphy.
  Interventions: Dietary Supplement: White chocolate mousse

INTERVENTIONS:
Dietary Supplement: Dark chocolate bar — Dark chocolate bar (70% cocoa solids (~500kcal, ~50% fat)), 100g / day for 3 days to assess postprandial brain activity and colonic transit by FDG-PET.
  Arms: Dark chocolate: FDG-PET
Dietary Supplement: Dark chocolate mousse — Dark chocolate mousse (150g, ~500kcal, ~50% fat) to assess gastric emptying and oro-caecal transit time by scintigraphy.
  Arms: Dark chocolate: Physiological Measurement
Dietary Supplement: White chocolate bar — White chocolate bar (0% cocoa solids (~500kcal, 50% fat)), 100g / day for 3 days to assess postprandial brain activity and colonic transit by FDG-PET.
  Arms: White chocolate: FDG-PET
Dietary Supplement: White chocolate mousse — White chocolate mousse (150g, ~500kcal, ~50% fat) to assess gastric emptying and oro-caecal transit time by scintigraphy.
  Arms: White chocolate: Physiological Measurement

SUMMARY:
This is a randomized, controlled, 2x2 cross-over study to assess the effects of cocoa solids on gastrointestinal transit, post-prandial sensation and well-being. Additionally functional brain imaging will be applied to identify regions of brain that are activated or inactivated by cocoa ingestion. Healthy subjects will be recruited and randomized to receive either dark chocolate (70% cocoa solids) or white chocolate (0% cocoa solids) in addition to their normal diet in randomized order. Reference standard methodology will be applied to measure gastric emptying, oro-caecal and colonic transit time. Dark and white chocolate (100g, ~500kcal, ~50% fat) will be consumed with radio-opaque markers on three consecutive days. On the third day chocolate ingestion will be followed by measurements of postprandial brain activity using FDG-Positron Emission Tomography. Additionally colonic transit will be assessed based on the number and distribution of radio-opaque markers in the colon. On the fourth day gastric emptying and oro-caecal transit time will be assessed by scintigraphy after ingestion of a dark or white chocolate mousse test meal (both 150g, ~500kcal, ~50% fat). During both interventional studies pre- and post-prandial satiety and dyspeptic symptoms, well-being and mood will be recorded. Additionally, validated questionnaires will assess digestive comfort and well-bring at the end of each study day. These results will deliver comprehensive information about the effects of cocoa on gastrointestinal transit and sensation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men and women)
* aged 18-65 years
* body mass index 18-30kg/m2.

Exclusion Criteria:

* special dietary requirements incompatible with dietary intervention (food allergies or intolerances)
* clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.) that preclude intake of test meals
* participation in another study with investigational drug within the 30 days preceding and during the present study (purely diagnostic studies are acceptable)
* individuals unwilling to provide written informed consent
* inability to follow the procedures of the study, e.g. due to language problems (all study documents in English)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-01; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Gastric emptying half time | Baseline until 2 hours postingestion
  assessed by scintigraphy

SECONDARY OUTCOMES:
Oro-caecal transit time (OCTT) | Baseline until 3 hours postingestion
  assessed by scintigraphy and 13-C Lactose-Ureide
Colonic transit time | Baseline until 3 days after ingestion
  assessed by radio-opaque marker technique
Post-prandial satiety | changes from baseline to three hours after treatment
  assessed by visual analogue scales
Gastrointestinal well-being | changes from baseline to three hours after treatment
  assessed by Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fox, Prof. Dr., Principal Investigator — St. Claraspital Basel, Abdominal Center: Gastroenterology
Locations (1):
- St Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided